CLINICAL TRIAL: NCT03360032
Title: A Comparative Assessment of Measurements Made in an Incremental Shuttle Walk Test and Incremental Cycle Ergometry Test in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Comparing Measurements Made in an Incremental Shuttle Walk Test and a Cardiopulmonary Exercise Test in Patients With IPF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 222072
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Incremental shuttle walk test; Cardiopulmonary exercise test; VO2 peak
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All patients will be asked to undertake an incremental shuttle walk test and a cardiopulmonary exercise test and the results will be compared.

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a chronic and potentially fatal lung disease. As IPF progresses, patients become increasingly breathless with reduced exercise capacity and quality of life. A cardiopulmonary exercise test (CPET) is a gold standard way of assessing patients with IPF.

An incremental shuttle walk test is simpler, cheaper, more widely available and anecdotally preferable to CPET. The investigators will compare the measurements made in an ISWT and a CPET in patients with IPF . We aim to determine whether sufficient information can be gathered in an ISWT to negate the need to undertake CPET.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a chronic and potentially fatal lung disease. As IPF progresses, patients become increasingly breathless with reduced exercise capacity and quality of life. Average life expectancy is three years from diagnosis but IPF progresses at different rates in different people. In 2012 the British Lung Foundation estimated that 32,500 in the UK had IPF.

An accurate prognosis can help determine the most appropriate individual treatment option and allow patients and their families to make suitable plans. Currently, measurements from resting lung function tests are used to predict prognosis. However, measurement made during CPET are more sensitive survival predictors and CPET is the gold standard test to assess prognosis in IPF. A CPET test is relatively time-consuming and requires specialist equipment that is not universally available. CPET is not routinely used in clinical practice for the assessment of IPF.

The incremental shuttle walk test (ISWT) is quicker, cheaper and more widely available than CPET. This study builds on previous research done by the Respiratory team which showed a linear relationship between the distance walked in an ISWT and peak oxygen consumption during a CPET, a useful prognostic predictor, in patients with interstitial lung disease. 40-50 patients with IPF will be recruited and will undertake both ISWT and CPET at University Hospital, Coventry. The investigators will compare the results in the current cohort to those of the previous study.

Additionally, the research team will compare oxygen pressure in capillary blood at the end of an ISWT and a CPET. The investigators will also compare patient experience of the two tests using questionnaires. This study paves the way for a simple, standardised test to more accurately predict prognosis in IPF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis confirmed by a multi-disciplinary team.
* Aged 16 or over
* Able to give informed consent to take part
* Able to undertake both a cycle ergometry test and an incremental shuttle walk test without needing walking aids

Exclusion Criteria:

* An inability to give informed consent.
* Taking part in a research project with a potentially research-modifying intervention
* Currently pregnant.
* Currently breastfeeding.
* Unable to perform an incremental shuttle walk test.
* Unable to perform an incremental cycle ergometry test.
* Unable to walk without an aid such as a stick or frame.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of idiopathic pulmonary fibrosis who are under the care of the Respiratory team at University Hospitals Coventry and Warwickshire NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
VO2 peak | Measured and reported at time of test
  Maximum oxygen consumption at peak exercise

SECONDARY OUTCOMES:
PO2 | Measured and reported at time of test
  Oxygen pressure in capillary blood at peak exercise

CONTACTS AND LOCATIONS:
Overall Officials: David Parr, Principal Investigator — University Hospitals Coventry and Warwickshire NHS Trust
Locations (1):
- University Hospital, Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT03360032/Prot_SAP_000.pdf